CLINICAL TRIAL: NCT00069628
Title: DirecNet Randomized Clinical Trial to Assess the Effectiveness of the GlucoWatch Biographer in the Management of Type 1 Diabetes in Children
Brief Title: Randomized Clinical Trial to Assess the Effectiveness of the GlucoWatch Biographer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: DirecNet 004; HD041890; HD041919-01; HD041908-01; HD041906-01; HD041918-01; HD041915
Record Dates: First submitted 2003-09-29; First posted 2003-09-30 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus, Insulin-Dependent
Keywords: Diabetes Mellitus, Insulin-Dependent; Type 1 Diabetes; Diabetes in Children; Continuous Glucose Monitoring Devices
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Continuous Glucose Monitoring

INTERVENTIONS:
Device: GlucoWatch® G2™ Biographer (GW2B)
Device: Continuous Glucose Monitoring System (CGMS)

SUMMARY:
This study will evaluate the safety and effectiveness of a continuous glucose monitor in children with Type 1 diabetes mellitus (T1DM).

DETAILED DESCRIPTION:
Intensive control of blood glucose levels has been shown to substantially prevent or delay complications of T1DM in adolescents and adults. The major limitation to implementation of intensive glycemic control is hypoglycemia. Younger children may be at increased risk for hypoglycemia, and the risk/benefit ratio of intensive glycemic control may be less favorable in this population. The Diabetes Research in Children Network (DirecNet) was established to evaluate the feasibility and effectiveness of intensive glycemic control in children with T1DM.

This study is designed to evaluate glycemic control, hypoglycemia, and quality of life when using a GlucoWatch G2TM Biographer (GW2B) versus standard care. Children in the study will use the GW2B in their home environment in order to assess if the GW2B can help to safely lower blood sugar levels (as measured by the glycosylated hemoglobin test), to learn how using the GW2B affects the daily lives of children with diabetes, and to find out if there are any drawbacks to using the GlucoWatch.

As part of the study, participants in the intervention group will also use a second glucose monitoring device called the Continuous Glucose Monitoring System (CGMS). The CGMS will be inserted at baseline and at Months 3 and 6; it will be worn for three days after each visit. The CGMS will be used to measure changes in biochemical hypoglycemia.

Participants at five participating centers will include a total of 200 children and adolescents with type 1 diabetes. Of the 200 children, 100 will be randomized to wear the GW2B and 100 will be randomized to usual care without GW2B. Each patient will be provided with a personal computer for weekly downloading of data and completion of questionnaires regarding hypoglycemia. Phone contacts will be made with the patients after Weeks 1, 2, and 4, then every 4 weeks to review their diabetes management. At Months 3, 6, 9 and 12, a follow-up visit will be performed to measure HbA1c. The CGMS sensor will be inserted to assess hypoglycemia at baseline and Months 3 and 6. At the 6-month follow-up visit, psychosocial questionnaires will also be administered.

ELIGIBILITY:
Inclusion Criteria

* Clinical diagnosis of type 1 diabetes
* Insulin therapy (either a pump or at least 2 injections per day) for at least one year prior to study entry
* HbA1c between 7.0 and 11.0%
* Stable insulin regimen for the 2 months prior to study entry and no plans to switch the modality of insulin administration during the next 6 months (e.g., injection user switching to a pump, pump user switching to injections, or the addition of Lantus [Glargine] insulin)
* Agree to comply with study requirements, including the performance of at least 4 fingerstick glucose checks a day using a home glucose monitor
* Comprehend written English
* Female participants must not intend to become pregnant during the next 6 months
* Plan to remain in the area of the clinical center during the next 6 months

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200
Dates: Start 2003-07; Study Completion 2004-11

PRIMARY OUTCOMES:
HbA1c value obtained 6 months after randomization

SECONDARY OUTCOMES:
Number of hypoglycemic events during 6 months
Diabetes Worry Scale at 6 months
PedsQL Diabetes Module at 6 months
Diabetes Self Management Profile at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: William V Tamborlane, MD, Study Chair — Yale University
Locations (6):
- United States (6):
  - Division of Pediatric Endocrinology and Diabetes, Stanford University, Stanford, California
  - Barbara Davis Center for Childhood Diabetes, University of Colorado, Denver, Colorado
  - Department of Pediatrics, Yale University School of Medicine, New Haven, Connecticut
  - Nemours Children's Clinic, Jacksonville, Florida
  - Jaeb Center for Health Research, Tampa, Florida
  - Department of Pediatrics, University of Iowa Carver College of Medicine, Iowa City, Iowa

REFERENCES:
- [Background] Tansey MJ, Beck RW, Buckingham BA, Mauras N, Fiallo-Scharer R, Xing D, Killman C, Tamborlane WV, Ruedy KJ; Diabetes Research in Children Network (DirecNet) Study Group. Accuracy of the modified Continuous Glucose Monitoring System (CGMS) sensor in an outpatient setting: results from a diabetes research in children network (DirecNet) study. Diabetes Technol Ther. 2005 Feb;7(1):109-14. doi: 10.1089/dia.2005.7.109. PMID 15738708
- [Background] Tamborlane WV, Kollman C, Steffes MW, Ruedy KJ, Dongyuan X, Beck RW, Chase P, Fox LA, Wilson DM, Tsalikian E; Diabetes Research in Children Network (DirecNet) Study Group. Comparison of fingerstick hemoglobin A1c levels assayed by DCA 2000 with the DCCT/EDIC central laboratory assay: results of a Diabetes Research in Children Network (DirecNet) Study. Pediatr Diabetes. 2005 Mar;6(1):13-6. doi: 10.1111/j.1399-543X.2005.00088.x. PMID 15787896
- [Background] Chase HP, Beck R, Tamborlane W, Buckingham B, Mauras N, Tsalikian E, Wysocki T, Weinzimer S, Kollman C, Ruedy K, Xing D. A randomized multicenter trial comparing the GlucoWatch Biographer with standard glucose monitoring in children with type 1 diabetes. Diabetes Care. 2005 May;28(5):1101-6. doi: 10.2337/diacare.28.5.1101. PMID 15855573
- [Background] Fiallo-Scharer R; Diabetes Research in Children Network Study Group. Eight-point glucose testing versus the continuous glucose monitoring system in evaluation of glycemic control in type 1 diabetes. J Clin Endocrinol Metab. 2005 Jun;90(6):3387-91. doi: 10.1210/jc.2004-2510. Epub 2005 Mar 22. PMID 15784705
- [Background] Diabetes Research in Children Network (DirecNet) Study Group. Diabetes self-management profile for flexible insulin regimens: cross-sectional and longitudinal analysis of psychometric properties in a pediatric sample. Diabetes Care. 2005 Aug;28(8):2034-5. doi: 10.2337/diacare.28.8.2034. No abstract available. PMID 16043752
- [Background] Diabetes Research in Children Network (DirecNet) Study Group. Youth and parent satisfaction with clinical use of the GlucoWatch G2 Biographer in the management of pediatric type 1 diabetes. Diabetes Care. 2005 Aug;28(8):1929-35. doi: 10.2337/diacare.28.8.1929. PMID 16043734
- [Background] William Tamborlane, Dongyuan Xing, Michael Steffes, Craig Kollman, Katrina Ruedy, Roy Beck, Rosanna Fiallo-Scharer, Larry Fox, Darrell Wilson, Eva Tsalikian, and the Diabetes Research In Children Network (DirecNet) Study Group: Performance of the DCA2000 for Measurement of Hemoglobin A1c Levels in Children with T1DM in a DirecNet Outpatient Clinical Trial. Pediatr Res 2004; 55 (4 Pt 2):138A.
- [Background] Michael Tansey, Roy Beck, Bruce Buckingham, Nelly Mauras, Rosanna Fiallo-Scharer, Dongyuan Xing, Craig Kollman, William Tamborlane, Katrina Ruedy, and the Diabetes Research in Children Network (DirecNet) Study Group: A Comparison of the Original vs. Modified Continuous Glucose Monitoring System (CGMS) Sensor During Using Data from Two DirecNet Studies. Diabetes 2004; 53(Suppl 2):A465.
- [Background] Rosanna Fiallo-Scharer, Dongyuan Xing, Stuart Weinzimer, Bruce Buckingham, Nelly Mauras, Michael Tansey, Roy Beck, Katrina Ruedy, Craig Kollman, William Tamborlane, and the Diabetes Research in Children Network (DirecNet) Study Group: Utility of CGMS as a Measure of Glycemic Control in Children with Type 1 Diabetes (T1DM). Diabetes 2004; 53(Suppl 2):A67.
- [Background] Peter Chase, Dongyuan Xing, Stuart Weinzimer, Bruce Buckingham, Nelly Mauras, Michael Tansey, Roy Beck, Katrina Ruedy, Craig Kollman, William Tamborlane, and the Diabetes Research in Children Network (DirecNet) Study Group: Comparison of 8-point Glucose Testing with Glycemic Control in Children with Type 1 Diabetes (T1DM). Diabetes 2004; 53(Suppl 2):A600.
- [Background] Tim Wysocki, Dongyuan Xing, Rosanna Fiallo-Scharer, Elizabeth Doyle, Jennifer Block, Eva Tsalikian, Roy Beck, Katrina Ruedy, Craig Kollman, William Tamborlane, and the Diabetes Research in Children Network (DirecNet) Study Group: Diabetes Self-Management Profile-Revised for Conventional and Flexible Insulin Regimens. Diabetes 2004; 53(Suppl 2):A436.
- [Background] H. Peter Chase, Roy Beck, William Tamborlane, Bruce Buckingham, Nelly Mauras, Eva Tsalikian, Tim Wysocki, Stuart Weinzimer, Katrina Ruedy, Dongyuan Xing, and the Diabetes Research in Children Network (DirecNet) Study Group: Lack of Effectiveness of the GlucoWatch G2 Biographer in Altering Glycemic Control in Children with Type 1 Diabetes. Diabetes Technol Ther 2005; 7(2):370.
- [Background] Darrell Wilson, Rosanna Fiallo-Scharer, Dongyuan Xing, Tim Wyscoki, Jennifer Block, Stu Weinzimer, Craig Kollman, Roy Beck, Katrina Ruedy, William Tamborlane, and the Diabetes Research in Children Network (DirecNet) Study Group: Reliability of Two Indices of the Biologic Variability in Glycosylation among Children and Adolescents with T1DM. Diabetes 2005; 54(Suppl 1):A454.